CLINICAL TRIAL: NCT03045523
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study to Evaluate GLPG2222 in Ivacaftor-treated Subjects With Cystic Fibrosis Harbouring One F508del CFTR Mutation and a Second Gating (Class III) Mutation
Brief Title: A Study to Evaluate GLPG2222 in Ivacaftor-treated Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG2222-CL-201
Record Dates: First submitted 2017-01-26; First posted 2017-02-07 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — GLPG2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG2222 Dose 1 (Experimental)
  Interventions: Drug: GLPG2222 150 mg q.d.
- GLPG2222 Dose 2 (Experimental)
  Interventions: Drug: GLPG2222 300 mg q.d.
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG2222 150 mg q.d. — GLPG2222 150 mg administered as a ready-to-use oral suspension, once daily (q.d.) for 29 days
  Arms: GLPG2222 Dose 1
Drug: GLPG2222 300 mg q.d. — GLPG2222 300 mg administered as a ready-to-use oral suspension, once daily (q.d.) for 29 days
  Arms: GLPG2222 Dose 2
Drug: Placebo — Placebo administered as a ready-to-use oral suspension, once daily (q.d.) for 29 days
  Arms: Placebo

SUMMARY:
This clinical study is a phase IIa, multi-center, randomized, double-blind, placebo-controlled, parallel group study to evaluate two doses of orally administered GLPG2222 in adult subjects with a confirmed diagnosis of CF harbouring one F508del CFTR mutation and a second gating (class III) mutation and on stable treatment with ivacaftor.

Up to 35 evaluable subjects are planned to be included in the study. Eligible subjects must be on stable treatment with physician prescribed ivacaftor (Kalydeco®) for at least 28 days at the baseline visit. They will be randomized in a 2:2:1 ratio to receive one of two active doses of GLPG2222 (150 mg q.d. or 300 mg q.d.) or placebo q.d. administered for 29 days. Subjects will be in the study for a minimum of 6 weeks and a maximum of 10 weeks, from screening until the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥ 18 years of age, on the day of signing the Informed Consent Form (ICF).
2. A confirmed clinical diagnosis of CF.
3. One F508del mutation on one allele in the CFTR gene, a gating (class III) mutation (one of the following: G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, or S549R) on the 2nd allele in the CFTR gene (documented in the subject's medical record or CF registry).
4. Weight ≥ 40 kg.
5. Stable concomitant treatment for at least 4 weeks (28 days) prior to baseline (including physician prescribed ivacaftor (Kalydeco®) 150 mg b.i.d.).
6. Forced expiratory volume in 1 second (FEV1) ≥ 40% of predicted normal for age, gender and height at screening (pre- or postbronchodilator).

Exclusion Criteria:

1. History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
2. Unstable pulmonary status or respiratory tract infection (including rhinosinusitis) requiring a change in therapy within 4 weeks of baseline.
3. Need for supplemental oxygen during the day, and >2 liters per minute (LPM) while sleeping.
4. History of hepatic cirrhosis with portal hypertension (e.g., signs/symptoms of splenomegaly, esophageal varices, etc).
5. Abnormal liver function test at screening; defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or alkaline phosphatase and/or total bilirubin (>1.5 times ULN (CTCAE Grade 2) and/or gamma-glutamyl transferase (GGT) ≥ 3x the upper limit of normal (ULN), and/or total bilirubin (>1.5 times ULN (CTCAE Grade 2).
6. Estimated creatinine clearance < 60mL/min using the Cockroft-Gault formula at screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Changes in adverse events | at screening and at each study visit up to day 43 which is the final FU visit
  To evaluate the safety and tolerability of GLPG2222 as compared to placebo in terms of adverse events
Changes in abnormal laboratory | at screening and at each study visit up to day 43 which is the final FU visit
  To evaluate the safety and tolerability of GLPG2222 as compared to placebo in terms of laboratory
Changes in abnormal vital signs, ECG or physical examination | at screening and at each study visit up to day 43 which is the final FU visit
  To evaluate the safety and tolerability of GLPG2222 as compared to placebo in terms of vital signs, ECG or physical examination

SECONDARY OUTCOMES:
Change from baseline of Sweat chloride concentration | at screening and at each study visit up to day 43 which is the final FU visit
Change from baseline of FEV1 (L) and percent predicted FEV1 for age, gender and height as assessed by spirometry | at screening and at each study visit up to day 43 which is the final FU visit
Change from baseline on the respiratory domain of Revised Cystic Fibrosis Questionnaire (CFQ-R) | at screening and at each study visit up to day 43 which is the final FU visit

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van Steen, MD, MBA, Study Director — Galapagos NV
Locations (22):
- Australia (4):
  - The Prince Charles Hospital, Chermside
  - The Alfred, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Westmead Hospital, Westmead
- Belgium (3):
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Fakultni nemocnice v Motole, Prague, Czechia
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - University Children´s Hospital, Tübingen
- Ireland (3):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St Vincents University Hospital, Dublin
- United Kingdom (8):
  - Birmingham Heartlands, Birmingham
  - Royal Devon and Exeter, Exeter
  - St James's University, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton Hospital, London
  - University Hospital of South Manchester, Manchester
  - Royal Victoria Infirmary, Newcastle
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Bell SC, Barry PJ, De Boeck K, Drevinek P, Elborn JS, Plant BJ, Minic P, Van Braeckel E, Verhulst S, Muller K, Kanters D, Bellaire S, de Kock H, Geller DE, Conrath K, Van de Steen O, van der Ent K. CFTR activity is enhanced by the novel corrector GLPG2222, given with and without ivacaftor in two randomized trials. J Cyst Fibros. 2019 Sep;18(5):700-707. doi: 10.1016/j.jcf.2019.04.014. Epub 2019 May 3. PMID 31056441